CLINICAL TRIAL: NCT01496196
Title: The Role of Inhalations of Tranexamic Acid in Patients With Hemoptysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0096-11-MMC
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2011-12

CONDITIONS: Hemoptisis
Keywords: hemoptisis; bleeding; tranexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tranexamic acid-500 mg/5 ml 3-4 times a day (Active Comparator): tranexamic acid arm: inhalations of tranexamic acid 500 mg/5 ml 3-4 times a day
  Interventions: Drug: tranexamic acid
- tranexamic (Placebo Comparator): placebo arm
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — 500 mg/5 ml 3-4 times a day
  Arms: tranexamic acid-500 mg/5 ml 3-4 times a day
Drug: tranexamic acid — 500 mg/5 ml 3-4 times a day
  Arms: tranexamic

SUMMARY:
Hemoptysis is defined as the expectoration of blood from respiratory tract, a spectrum that varies from blood-streaking of sputum to coughing up large amounts of pure blood.

Massive hemoptysis variably defined as the expectoration of 100-600 ml over 24-h period.

The most common site of bleeding is the tracheobronchial tree, which can be affected by inflammation (acute or chronic bronchitis, bronchiectasis) or by neoplasm ( bronchogenic carcinoma, endobronchial metastatic carcinoma, bronchial carcinoid tumor). The bronchial arteries, which originate either from aorta or from intercostal arteries, and are part of the high-pressure systemic circulation, are the source of bleeding in bronchitis or bronchiectasis or endo bronchial tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Hemodynamicaly stable
* Hemoptysis of varying etiologies
* Coumadin treatment will be switched to clexane or heparine

Exclusion Criteria:

* Age < 18
* Hemodinamicaly unstable
* Massive hemoptysis ( > 200 ml / day)
* Renal failure: creatinine > 3, renal replacement treatment
* Hepatic failure: bilirubin > 2 mg/dl, AST > 3 of upper normal limit level
* Coagulation disorders, INR> 2.
* Hypesensitivity to tranexamic acid
* Pregnant woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
bleeding stops | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, Dr., Principal Investigator — Meir Medical Center, Kfar Saba, Israel
Locations (1):
- Pulmonary department, Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Derived] Wand O, Guber E, Guber A, Epstein Shochet G, Israeli-Shani L, Shitrit D. Inhaled Tranexamic Acid for Hemoptysis Treatment: A Randomized Controlled Trial. Chest. 2018 Dec;154(6):1379-1384. doi: 10.1016/j.chest.2018.09.026. Epub 2018 Oct 12. PMID 30321510